CLINICAL TRIAL: NCT00202020
Title: Cilostazol Stroke Prevention Study-a Randomized, Double Blind, Double Dummy, Parallel Comparative, Multicenter Clinical Trial
Brief Title: Efficacy and Safety Study of Cilostazol to Prevent Reoccurrence of Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Collaborators: Zhejiang Otsuka Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OBRI0001
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-03-16 (Estimated); Status verified 2006-03

CONDITIONS: Cerebral Infarction
Keywords: Cerebral infarction; Prevention; Cilostazol; Aspirin; Stroke; Clinical trial
MeSH Terms: conditions — Cerebral Infarction; Stroke | interventions — Cilostazol; Aspirin

INTERVENTIONS:
Drug: Cilostazol 200mg/day Oral
Drug: Aspirin 100mg/day Oral

SUMMARY:
The study design is subject to relevant SFDA regulations about clinical trials. This indication was approved in Japan in 2003.

From the end of May 2004 to the end of Dec. 2004, 720 patients with previous cerebral infarction(see the inclusion criteria) were enrolled in to the study and received one of the two treatment regimens, Cilostazol or Aspirin, the ratio of patient number of each group is 1:1. For each patient, the chance of entering either of these two groups is the same. The treatment will continue till the end of 2005. During the treatment period, patients will be observed concerning some certain events, mainly reoccurrence of stroke. If the patient experiences reoccurrence of stroke, or other event that the doctors think it is not appropriate to continue the study medication, this patient would stop the treatment. Patients were also required to take MRI head scan before entering the study and on completion of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had cerebral infarction within 6 months and 1 month before entry 2. Within a few days of the onset of cerebral infarction onset, CT or MRI showed evidence of infarction that could be responsible for this stroke onset 3. A modified ranking scale of less than 4 4. Aged 18~75 5. Consent of the patients or their legal guardians

-

Exclusion Criteria:

1. History of intracranial hemorrhage 2. Stroke secondary to cardiogenic embolism 3. Serious damage of motorial function, dementia 4. Serious complications or co morbidity(uncontrolled accelerated type of hypertension, BP>180/120mmHg, diabetic acidosis, heart failure, renal failure, hepatocirrhosis, malignant tumor) 5. Contraindication of Cilostazol and Aspirin 6. Patients who need co medication of other antiplatelet agents, anticoagulants or fibrinolytic drugs 7. Active peptic ulcer 8. Pregnancy or breast feeding 9. Judged to be inappropriate to enter the study by investigators. -

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720
Dates: Start 2004-05; Study Completion 2006-01

PRIMARY OUTCOMES:
Recurrence of stroke(cerebral infarction/haemorrhage/subarachnoid haemorrhage)

SECONDARY OUTCOMES:
Recurrence of cerebral infarction detected in MRI
Death due to cerebral vascular events
Myocardial infarction
Vascular events(acute artery thrombosis/embolism, pneumonia embolism, venous thrombosis, angina pectoris)
TIA
Death

CONTACTS AND LOCATIONS:
Overall Officials: Yi N Huang, Professor, Principal Investigator — Peking University First Hospital
Locations (12):
- China (12):
  - 1st affiliated hospital, Guangzhou Zhongshan University, Guangzhou, Guangdong
  - 2nd affiliated hospital, Guangzhou medical college, Guangzhou, Guangdong
  - 1st affiliated Jilin University, Changchun, Jilin
  - 1st affiliated hospital, Xi'an Jiatong University, Xi’an, Shanxi
  - 2nd affiliated hospital, Zhejiang University, Hangzhou, Zhejiang
  - 1st affiliated hospital, Peking University, Beijing
  - 3rd affiliated hospital, Peking University, Beijing
  - General Hospital of Beijing Military Area of PLA, Beijing
  - Renmin Hospital, Peking University, Beijing
  - Huashan Hospital Shanghai Fudan University, Shanghai
  - Renji Hospital, Shanghai 2nd medical university, Shanghai
  - General Hospital, Tianjin Medical University, Tianjin

REFERENCES:
- [Derived] Liu W, Liu R, Sun W, Peng Q, Zhang W, Xu E, Cheng Y, Ding M, Li Y, Hong Z, Wu J, Zeng J, Yao C, Huang Y; CASISP Study Group. Different impacts of blood pressure variability on the progression of cerebral microbleeds and white matter lesions. Stroke. 2012 Nov;43(11):2916-22. doi: 10.1161/STROKEAHA.112.658369. Epub 2012 Sep 4. PMID 22949472
- [Derived] Huang Y, Cheng Y, Wu J, Li Y, Xu E, Hong Z, Li Z, Zhang W, Ding M, Gao X, Fan D, Zeng J, Wong K, Lu C, Xiao J, Yao C; Cilostazol versus Aspirin for Secondary Ischaemic Stroke Prevention cooperation investigators. Cilostazol as an alternative to aspirin after ischaemic stroke: a randomised, double-blind, pilot study. Lancet Neurol. 2008 Jun;7(6):494-9. doi: 10.1016/S1474-4422(08)70094-2. Epub 2008 May 2. PMID 18456558